CLINICAL TRIAL: NCT01960478
Title: Predictive Value of Copeptin in the Diagnosis of Acute Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5476
Record Dates: First submitted 2013-09-25; First posted 2013-10-10 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Vascular Accident (CVA)
MeSH Terms: conditions — Stroke | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bood test (Other)
  Interventions: Biological: (for each intervention); Other: Blood test

INTERVENTIONS:
Biological: (for each intervention)
Other: Blood test

SUMMARY:
In the USA, every year 795,000 patients suffer a cerebral vascular accident (CVA), which represents a yearly cost of $73.7 billion. CVA is the third main cause of death and the main source of acquired handicap in adults, as a result it is now a key priority in public health and part of " The CVA National Action Plan 2013-2014".

Copeptin is a polypeptide, by- product of Vasopressin metabolism. The increase of Copeptin plasma level, as for Vasopressin, is connected to hydric balance disorders found in cardio-vascular, renal and endocrine diseases. This link has already shown its interest in the early diagnosis of myocardial infarction and, in a more indirect way, CVA.

Copeptin is associated with acute endogenous stress. It seems to have interesting potential in the diagnosis of CVA by its negative predictive value like D-dimeres in pulmonary embolism. Proadrenomedullin and Brain Natriuretic Peptide (BNP) are both associated with the prognosis of cardio-vascular diseases and could be interesting in evaluating CVA prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients, male or female, may be included if they meet the following criteria:
* patients with suspected ischemic CVA admitted in an acute stroke unit (thrombolysis unit).
* aged 18 and over.
* MRI Scan undertaken under the current protocol which includes the following sequences: distribution, T2* (gradient echo), ARM, TOF and FLAIR.
* after information given the consent form is signed:

  * by the patient .or for those unable to express their consent (in case of coma or severe neurological disorder) by a relative or next of kin.

.the patient will be informed as soon as he has recovered his faculties in order to be able to express, if he wishes, his opposition to the pursuit of the research (sample destruction before tested).

- the patient must be registered with the Social Security

Exclusion Criteria:

All patients with a contraindication to MRI Scan:

* Pacemaker,
* Implanted cardiac defibrillator,
* Implanted Neuro-stimulator,
* Cochlear Implants
* Implanted Insulin pump
* Other implanted electronic medical device
* Vascular intracerebral Clip
* Cardiac Valve
* Other metallic implant
* Metallic foreign body
* Ventricular diversion valve
* Eye or hearing prosthesis
* Current or suspected pregnancy
* Breast feeding

Those who are under protection of justice, under guardianship or curatorship will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-01-07 (Actual); Primary Completion 2014-10-05 (Actual); Study Completion 2014-10-05 (Actual)

PRIMARY OUTCOMES:
Determine the minimum level of Copeptin required to determine if the patients present with acute CVA or not. | Participants will be followed during 90 days
  Copeptin is associated with acute endogenous stress. It seems to have interesting potential in the diagnosis of CVA by its negative predictive value like D-dimers in pulmonary embolism. Proadrenomedullin and Brain Natriuretic Peptide (BNP) are both associated with the prognosis of cardio-vascular diseases and could be interesting in evaluating CVA prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien HARSCOAT, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service des Urgences Médico-Chirugicales Adultes Hôpitaux Universitaires, Strasbourg, France